CLINICAL TRIAL: NCT01012856
Title: Explicit and Implicit Change of Depression in Exposure-based Cognitive Therapy
Brief Title: Randomized Clinical Trial of an Exposure-based Cognitive Therapy for Depression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PP00P1_ 123377
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Unipolar Depression
Keywords: depressive episode; psychotherapy; cognitive therapy; emotional processing; RCT; exposure; dual process model; Implicit Association Test; mechanism of change
MeSH Terms: conditions — Depressive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-Behavioral Therapy for Depression (CBT) (Active Comparator)
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Depression
- Exposure-Based Cognitive Therapy for Depression (EBCT) (Experimental)
  Interventions: Behavioral: Exposure-Based Cognitive Therapy for Depression

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy for Depression — 22 weekly sessions and 2 booster session of face to face outpatient psychotherapy; focus on cognitive restructuring without emotion-focused interventions
  Arms: Cognitive-Behavioral Therapy for Depression (CBT)
Behavioral: Exposure-Based Cognitive Therapy for Depression — 22 weekly sessions and 2 booster session of face to face outpatient psychotherapy; focus on emotion-focused interventions
  Arms: Exposure-Based Cognitive Therapy for Depression (EBCT)

SUMMARY:
The purpose of this study is to investigate, if exposure-based cognitive therapy (EBCT) is at least as effective as the established cognitive-behavioral therapy and more effective in its long-term efficacy. Moreover the mechanisms of change of the EBCT are investigated.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder according to DSM-IV as main diagnosis
* minimum standardized depression scores (BDI >= 17; HAMD >=13)
* minimum age of 18 years
* informed consent to participate voluntarily in the study
* sufficient German language skills

Exclusion Criteria:

* acute suicidality
* depressive disorder with mood-incongruent psychotic features
* chronic depressive disorder
* organic cause of depression
* drug-induced depression
* bipolar disorder
* diagnosis of schizophrenia, schizophreniform, schizoaffective disorders, and/or psychosis NOS
* comorbid dysthymia, psychotic disorder (acute or anamnestic), dementia, substance dependence, schizotypal/ borderline/ or antisocial personality disorder
* psychopharmacological treatment other than antidepressants
* antidepressant medication, if it is changed within one month prior to the beginning of psychotherapy
* other simultaneous psychological treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
severity of depressive symptoms measured by the Beck-Depression-Inventory (BDI-II) | end of therapy, 6 month after end of therapy (follow up)

SECONDARY OUTCOMES:
symptom impairment measured by the Brief Symptom Inventory (BSI) | end of therapy, 6-month follow up
quality of life measured by the WHO Quality of Life-BREF (WHOQOL-BREF) | end of therapy, 6-month follow-up
interpersonal problems measured by the Inventory of Interpersonal Problems (IIP) | end of therapy, 6-month follow-up
avoidance measured by the Cognitive-Behavioral Avoidance Scales (CBAS) | end of therapy, 6-month follow-up
resources measured by the Bernese Inventory of Resources (RES-K) | end of therapy, 6-month follow-up
explicit self-esteem measured by the Rosenberg self-esteem scale (RSES) | end of therapy, 6-month follow up
implicit self-esteem measured by the Self-Esteem Implicit Association Test (SE-IAT) | end of therapy
goal attainment measured by Goal Attainment Scaling (GAS) | end of therapy
avoidance motivation measured by the Inventory of Approach and Avoidance Motivation (IAAM) | end of therpy, 6-month follow-up
motivational incongruence measured by The Incongruence Questionnaire (INC) | end of therapy, 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Martin Grosse Holtforth, Professor MD, Principal Investigator — University of Zurich, Department of Psychology
Locations (1):
- University of Zurich, Department of Psychology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Hayes AM, Feldman GC, Beevers CG, Laurenceau JP, Cardaciotto L, Lewis-Smith J. Discontinuities and cognitive changes in an exposure-based cognitive therapy for depression. J Consult Clin Psychol. 2007 Jun;75(3):409-421. doi: 10.1037/0022-006X.75.3.409. PMID 17563158
- [Background] Hayes AM, Strauss JL. Dynamic systems theory as a paradigm for the study of change in psychotherapy: an application to cognitive therapy for depression. J Consult Clin Psychol. 1998 Dec;66(6):939-47. doi: 10.1037//0022-006x.66.6.939. PMID 9874907
- [Background] Hayes AM, Laurenceau JP, Feldman G, Strauss JL, Cardaciotto L. Change is not always linear: the study of nonlinear and discontinuous patterns of change in psychotherapy. Clin Psychol Rev. 2007 Jul;27(6):715-23. doi: 10.1016/j.cpr.2007.01.008. Epub 2007 Jan 19. PMID 17316941
- [Background] Beevers CG. Cognitive vulnerability to depression: a dual process model. Clin Psychol Rev. 2005 Nov;25(7):975-1002. doi: 10.1016/j.cpr.2005.03.003. PMID 15905008
- [Background] Pascual-Leone A. Dynamic emotional processing in experiential therapy: two steps forward, one step back. J Consult Clin Psychol. 2009 Feb;77(1):113-26. doi: 10.1037/a0014488. PMID 19170458
- [Derived] Babl A, Rubel J, Gomez Penedo JM, Berger T, Grosse Holtforth M, Eubanks CF. Can session-by-session changes in self-reported alliance scores serve as a measure of ruptures in the therapeutic alliance? J Consult Clin Psychol. 2024 Feb;92(2):129-133. doi: 10.1037/ccp0000861. Epub 2023 Nov 27. PMID 38010758
- [Derived] Grosse Holtforth M, Krieger T, Zimmermann J, Altenstein-Yamanaka D, Dorig N, Meisch L, Hayes AM. A randomized-controlled trial of cognitive-behavioral therapy for depression with integrated techniques from emotion-focused and exposure therapies. Psychother Res. 2019 Jan;29(1):30-44. doi: 10.1080/10503307.2017.1397796. Epub 2017 Nov 12. PMID 29130400